CLINICAL TRIAL: NCT01525160
Title: Novel Biomarkers for Haemostasis in Patients With the Obstructive Sleep Apnoea Hypopnoea Syndrome
Brief Title: New Markers to Measure Clotting in Patients With the Obstructive Sleep Apnoea Hypopnoea Syndrome
Status: Completed | Type: Observational
Sponsor: Hywel Dda Health Board (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Abertawe Bro Morgannwg University NHS Trust (Other Government); Swansea University (Other)
Responsible Party: Principal Investigator, Dr Maria Wilczynska, Clinical Research Fellow in Respiratory Medicine, Hywel Dda Health Board
Other Study IDs: RES-54
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Obstructive Sleep Apnoea Hypopnoea Syndrome; Biomarkers of Fibrin Clot Structure; Biomarkers of Vascular Endothelial Injury
Keywords: Clot structure; Haemostasis; Gel point; Fractal dimension; serum amyloid A; C-reactive protein; vascular cell adhesion molecule-1; intercellular adhesion molecule-1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen aliquots of citrated plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Obstructive Sleep Apnoea Hypopnoea Syndrome(OSAHS)affects at least 4% of males and 2% of females.

OSAHS is the combination of excessive daytime sleepiness, snoring and apnoeas (stopping breathing at night). As well as affecting tiredness, mood, concentration and quality of life - there is growing concern that it can increase the risk of high blood pressure, heart problems, strokes and thromboses (clots in the veins).

It appears that OSAHS may affect the thickness of the blood and cause it to clot more easily it also causes damage to the lining of the blood vessels (endothelial injury). These effects seem independent of other risk factors such as obesity, smoking, family history of clots etc.

The investigators are testing new biomarkers: gel point and fractal dimension developed at the Swansea University to measure the 'clotting' of the blood in people with OSAHS and a similar group of people who snore and who are sleepy but do not have OSAHS on sleep studies (Controls) Also markers of vascular inflammation are being measured.

DETAILED DESCRIPTION:
Primary objective:

The primary outcome of this study is to test the null hypothesis that no significant difference exists between fractal dimension (Df)and vascular injury markers including serum amyloid A (SAA), C-reactive protein (CRP), vascular cell adhesion molecule-1 (VCAM-1) and intercellular adhesion molecule-1 (ICAM-1)in patients with OSAHS and sleepy, snoring controls of similar age, gender and BMI.

Secondary objectives:

1. To test the null hypothesis that there is no significant difference in measured markers before and after a night's sleep in OSAHS and controls.
2. To test the null hypothesis that there is no significant difference in measured markers following 1 month of CPAP treatment, in those with OSAHS.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 year old with h/o daytime sleepiness, snoring and apnoeas

Exclusion Criteria:

* Refusal to give written informed consent.
* Personal or family history of pro- thrombotic or bleeding disorders, severe liver disease (clotting problems) and those prescribed warfarin or heparin.
* Those with borderline sleep studies (4% Diprate or AHI 10-14 per hour).
* Aged less than 18 years or greater than 80 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are recruited prospectively from a specialist sleep-disordered breathing clinic in Prince Philip Hospital, Hywel Dda Health Board. They are referred from both primary and secondary care with varying degrees of symptoms suggestive of OSAHS (daytime sleepiness, snoring and/or nocturnal apneas).
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Difference between fractal dimension (Df) in patients with OSAHS and controls | 18 months

SECONDARY OUTCOMES:
Difference in Df before and after a night's sleep in OSAHS and controls. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Kier Lewis, MD MBChB, Principal Investigator — Prince Philip Hospital; Phillip A Evans, Prof, Study Director — Morriston Hospital
Locations (1):
- Prince Philip Hospital, Llanelli, Dafan, United Kingdom